CLINICAL TRIAL: NCT05893966
Title: Prospective Cohort for Tumor Bed Boost Radiotherapy in HER2 Positive Breast Cancer
Acronym: BOOST-HER2
Status: Recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Haeyoung Kim, Associate professor, Samsung Medical Center
Other Study IDs: 2022-11-018
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Whole breast irradiation +/- tumor bed boost — Postoperative whole breast irradiation (3D-conformal radiation therapy or IMRT) with or without tumor bed boost (sequential or simultaneous integrated boost)

SUMMARY:
The purpose of this study is to analyze treatment outcomes related to tumor bed boost of postoperative radiation therapy in patient with HER2+ breast cancer who underwent breast conserving surgery.

The main questions it aims to answer are:

* 7-year ipsilateral breast tumor recurrence
* 7-year disease-free survival
* 7-year locoregional recurrence
* 7-year overall survival
* Adverse events of radiation therapy

Participants will be assessed by multi-dimensional methods after radiation therapy:

* Assessment for the disease status (disease-free or recurrence) including physical and radiologic examination
* Assessment for the adverse events according to CTCAE version 5.0

ELIGIBILITY:
Inclusion Criteria:

* Female patients with age minimum 19
* Pathological confirmation of HER2+ invasive breast cancer
* Eastern Cooperative Oncology Group performance status 0-2
* Informed consent of the participant

Exclusion Criteria:

* Pathological confirmation of ductal carcinoma in situ of the breast
* Previous history of radiation therapy to ipsilateral breast

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any HER2+ invasive breast cancer patient with eligible performance except previous history of radiation therapy to ipsilateral breast
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-11-29 (Actual); Primary Completion 2025-11-29 (Estimated); Study Completion 2032-11-29 (Estimated)

PRIMARY OUTCOMES:
Ipsilateral breast tumor recurrence | 7 years from the start of the postoperative radiation therapy
  The event for ipsilateral breast tumor recurrence (IBTR) was defined as any breast tumor recurrence in irradiated breast.

SECONDARY OUTCOMES:
Disease-free survival | 7 years from the start of the postoperative radiation therapy
  The event for disease-free survival (DFS) was defined as any local, regional, or distant recurrence or breast cancer-related death.
Locoregional recurrence | 7 years from the start of the postoperative radiation therapy
  The event for locoregional recurrence was defined as recurrence in irradiated breast / chest wall or regional lymph node area.
Overall survival | 7 years from the start of the postoperative radiation therapy
  The event for overall survival (OS) was defined as death of any cause.
Adverse events | 7 years from the start of the postoperative radiation therapy
  Adverse events were evaluated and graded according to CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Haeyoung Kim, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea